CLINICAL TRIAL: NCT06120855
Title: The Safer Cannabis - Research In Pharmacies Randomized Controlled Trial (SCRIPT)
Brief Title: Study on Regulated Cannabis Sales in Pharmacies
Acronym: SCRIPT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Universität Luzern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SCRIPT
Record Dates: First submitted 2023-10-19; First posted 2023-11-07 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Marijuana Smoking; Cannabis; Cannabis Use
Keywords: Cannabis; Cannabis Use; Cannabis sativa; Cannabinoids
MeSH Terms: conditions — Marijuana Smoking; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: This is a multicenter, pragmatic, open-labelled randomized controlled trial from baseline to 6-months follow-up. After 6 months, the control group is allowed to purchase cannabis in pharmacies, too, and the study design changes to a cohort-study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regulated cannabis from authorized pharmacies (intervention group) (Experimental): Multimodal intervention of authorized, regulated cannabis sale in combination with counselling on reducing harms for recreational cannabis users in Swiss pharmacies (intervention group).
  Interventions: Drug: Regulated cannabis from authorized pharmacies
- Cannabis from the illicit market (control group) (Active Comparator): The control group receives no intervention and is expected to continue purchasing cannabis from the illicit market.
  Interventions: Drug: Cannabis from the illicit market

INTERVENTIONS:
Drug: Regulated cannabis from authorized pharmacies — The intervention group is allowed to purchase regulated cannabis in authorized pharmacies. The intervention includes various offers: Participants can choose between cannabis sorts and delivery methods, and they are encouraged to shift from smoking cannabis to vaping cannabis-containing e-liquids, vaporizing cannabis blossoms or using oral cannabis. Vaping / vaporizing electronic devices are also recommended. At the same time, pharmacists offer opportunistic smoking cessation and problematic cannabis, alcohol use and further drug use counseling that conforms to motivational interviewing principles.
  Study participants can choose between different cannabis-containing products such as dried cannabis flowers, cannabis concentrates (colloquially called hashish or hash), e-liquids and oral cannabis. Besides the cannabis products, participants can buy vaping or vaporizing electronic devices at the pharmacy (they are not considered as study products).
  Arms: Regulated cannabis from authorized pharmacies (intervention group)
Drug: Cannabis from the illicit market — The control group receives no intervention and is expected to continue purchasing cannabis from the illicit market.
  Arms: Cannabis from the illicit market (control group)

SUMMARY:
Though regulated cannabis sales are increasing, little is known about the individual health effects of cannabis regulation. Data from countries with a regulated market can be used to test the effect of regulation on the price of cannabis in the illicit market, and to explore its effect on social and health outcomes at the societal level, but strength of evidence for individual health and social outcomes is more limited because it must be aggregated on a state or country level. Data on individual and social outcomes should include baseline measurements before and outcome measurements after regulations changed. In this context, randomized-controlled trials are the least biased source of data on the effects of interventions.

The SCRIPT study aims to investigate the individual health and social impact on recreational cannabis users who are allowed to purchase authorized, regulated cannabis from Swiss pharmacies compared to users who buy cannabis on the illicit market. Participants are randomly allocated in one of the two groups and followed-up for 6 months. After 6 months, all participants are allowed to participate in the intervention and the cohort is followed up for another 18 months.

The intervention includes various offers: Participants can choose between cannabis sorts and delivery methods, and they are encouraged to shift from smoking cannabis to vaping cannabis-containing e-liquids, vaporizing cannabis blossoms or using oral cannabis. Vaping / vaporizing electronic devices are also recommended. At the same time, pharmacists offer opportunistic smoking cessation and problematic cannabis, alcohol use and further drug use counseling that conforms to motivational interviewing principles.

The SCRIPT study adheres to rigorous quality criteria for the production and storage of regulated cannabis products. Only vaping / vaporizing electronic devices which are validated to reduce exposure to toxicants compared to cannabis smoking are recommended.

DETAILED DESCRIPTION:
Cannabis is the most consumed illegal substance in Switzerland. Many countries and an increasing number of US states have regularized cannabis production and distribution for non-medical use. Analyses of the effects of regulation are promising on a population level, but the causal effects of regulation have only been assessed in before-after studies or ecological comparisons between countries or states. Randomized controlled trials (RCT) are needed to better assess the effects of cannabis regulation on individuals. Since May 2021, the conduct of scientific pilot studies are allowed in Switzerland. While rigorous quality and safety standards cannot be implemented in illicit production and distribution networks, they can be implemented in regulated markets. Beyond psychiatric outcomes, the major hazard associated with cannabis use on somatic health outcomes are mostly related to smoking cannabis and mixing it with tobacco. Regulation therefore also opens the door to harm reduction strategies like counseling users to vape, vaporize, or eat cannabis instead of smoking it. Regulated sale in pharmacies would further facilitate smoking cessation counseling and access to health and social care for those in need. The SCRIPT trial aims to investigate the individual health and social impact on recreational cannabis users who are offered a multimodal intervention of authorized, regulated cannabis sale in combination with counselling on reducing harm (intervention group) compared to users who continue to buy cannabis on the illicit market (control group).

The intervention group is allowed to purchase regulated cannabis in authorized pharmacies. The intervention includes various offers: Participants can choose between cannabis sorts and delivery methods, and they are encouraged to shift from smoking cannabis to vaping cannabis-containing e-liquids, vaporizing cannabis blossoms or using oral cannabis. Vaping / vaporizing electronic devices are also recommended. At the same time, pharmacists offer opportunistic smoking cessation and problematic cannabis, alcohol use and further drug use counseling that conforms to motivational interviewing principles. The control group receives no intervention and is expected to continue purchasing cannabis from the illicit market.

This is a multicenter, pragmatic, open-labelled randomized controlled trial from baseline to 6-months follow-up. After 6 months, the control group is allowed to purchase cannabis in pharmacies, too, and the study designs changes to a cohort-study.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old (validated with valid identification document)
* Written informed consent
* Regular cannabis user: Self-reported cannabis use at least once a month over the last 6 months and verified cannabis exposure based on urine analysis at baseline
* Resident status in the canton of Bern (for cannabis purchase in the cities of Bern or Biel) or in the city of Lucerne (for cannabis purchase in the city of Lucerne) (validated with registration confirmation from the municipality or confirmation of the residential address)

Exclusion Criteria:

* Pregnant women (pregnancy test based on urine sample)
* Breastfeeding women (self-reported)
* People with a prescription for medical cannabis (self-reported)
* People currently in psychiatric inpatient treatment (self-reported)
* People with current, severe psychosis (self-reported and confirmed by study nurse/study physician)
* People with current, severe suicidal thoughts (self-reported and confirmed by study nurse/study physician)
* Inability to follow the procedures of the study due to severe cognitive impairment or language problems
* People who cannot attend the baseline study visit in-person
* People planning to move out of the canton of residence within 6 months of entering the trial.
* People who are participating or have participated (inclusion date up to one year ago) in another cannabis pilot trial which allows to buy regulated cannabis (validated by matching untraceable codes between studies witch the same catchment area).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1091 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-03-11 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Self-reported cannabis and tobacco smoking abstinence in the 7 days prior to the 6-months follow-up visit, validated by carbon monoxide (CO) in exhaled air | 6 months
  To distinguish between non-smoker and smoker, the cut-off for the CO measurement is <10 parts per million (ppm) and no self-reported combustible cannabis and tobacco use within the last 7 days (7-day point prevalence of abstinence). The validation is based on the worst-case principle. Smokers are considered as
  * participants with a positive CO measurement, even if the self-report is negative.
  * participants with a positive self-declaration, even if the CO measurement is negative.

SECONDARY OUTCOMES:
Self-reported reported 7-days point prevalence abstinence from cannabis and tobacco smoking at 6 months follow-up, without validation by CO in exhaled air. | 12, 18, & 24 months
  Based on interviews by phone or online
Shift from smoking to safer, alternative delivery methods of cannabis and, if applicable, tobacco. | 6, 12, 18, & 24 months
  Shift from smoking cannabis to safer, alternative delivery methods of cannabis and, if applicable, from smoking tobacco to alternative nicotine delivery systems or nicotine cessation between groups among those who were smoking cannabis at baseline and/or were smoking tobacco at baseline, with and without validation
Concentration of toxicants in urine | 6 months
  Measured in urine from a sub-sample
Type of cannabis sold per participant in pharmacies | 6, 12, 18, & 24 months
Amount of cannabis sold per participant in pharmacies | 6, 12, 18, & 24 months
Self-reported cannabis purchase on the illicit market | 6, 12, 18, & 24 months
Self-reported frequency of use | 6, 12, 18, & 24 months
Concentration of THC and CBD in cannabis bought on the illicit market | 6 months
  Measured in cannabis from a random sub-sample.
Concentration of contaminants in cannabis bought on the illicit market | 6 months
  Measured in cannabis from a random sub-sample.
Severity of generalised anxiety disorder | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome. Measured by Generalised Anxiety Disorder (GAD-7) questionnaire (scores range from 0 to 21, with higher scores indicating higher levels of generalised anxiety)
Attention Deficit Hyperactivity Disorder (ADHD) symptoms in adults | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome. Measured by Adult ADHD Self-Report Scale (ASRS) questionnaire.
Severity of depression | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome. Measured by the Patient Health Questionnaire-9 (PHQ-9) (scores range from 0 to 27, with higher scores indicating more depressive symptoms)
Number of psychotic symptoms | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome. Measured by the Psychotic Symptoms (PS) Checklist
Somatic health | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome. Measured by Pittsburgh Sleep Quality Index (PSQ-I) questionnaire.
Impact of COPD | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome. Measured by COPD Assessment Test (CAT) questionnaire (scores range from 0 to 40, with higher scores indicating indicating a more severe impact of COPD on a patient's life).
Severity of dyspnea | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome. Measured by Modified Medical Research Council (MMRC) scale for dyspnea.
COPD exacerbation assessment | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome.
Quality of life (health-related) | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome. Measured by the European Quality of Life-5 Dimensions (EQ-5D) questionnaire.
Perception of stress | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome. Measured by the Perceived Stress Scale (PSS).
Cannabis use and purchase behavior | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome.
Cannabis use disorder | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome. Measured by Cannabis Use Disorders Identification Test - Revised (CUDIT-R) questionnaire.
Consumption motives | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome.
Consumption competence | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome.
Consumption risk perception | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome.
Nicotine/tobacco use behavior | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome
Exposure to second-hand smoke | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome
Alcohol consumption behavior | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome. Measured by Alcohol Use Disorders Identification Test (AUDIT-C).
Drug consumption behavior | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome. Measured by Alcohol, Smoking and Substance Involvement Screening Test (ASSIST V3.0).
Medication use behavior | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome
Treatment/Counseling Experience | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome
Use of health and social services | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome.
Body mass index | 6 months
  Cardiovascular risk factor (CVRF) measured at physical examinations.
Blood pressure | 6 months
  Cardiovascular risk factor (CVRF) measured at physical examinations.
Waist-to-hip ratio | 6 months
  Cardiovascular risk factor (CVRF) measured at physical examinations.
Number of safety events | 6, 12, 18, & 24 months
  Recorded as participant-reported outcome.
Inflammation-related protein biomarkers | 6 months
  Measured from blood samples from a sub-sample. Analysis of 92 protein biomarkers associated with inflammatory and immune response processes using the Olink® Target 96 Inflammation Panels.
Blood biomarker for alcohol and cannabis exposure | 6 months
  Validation of the self-reported exposure to alcohol and cannabis through biomarkers of exposure, measured from blood samples from a sub-sample

OTHER OUTCOMES:
Gene activity related to chronic cannabis use | Baseline
  The analysis of gene activity related to chronic cannabis use is exploratory; it is measured through epigenetic methylation from a blood sample collected from a sub-sample

CONTACTS AND LOCATIONS:
Overall Officials: Reto Auer, Prof., Study Chair — Institute of Primary Health Care (BIHAM), Faculty of Medicine, University of Bern
Locations (2):
- Switzerland (2):
  - University of Bern, Bern
  - Zentrum für Hausarztmedizin und Community Care, University of Lucerne, Lucerne

IPD SHARING:
Plan to Share IPD: No